CLINICAL TRIAL: NCT01204008
Title: A Prospective Randomized Trails for Primary Disc Herniation With Radiculopathy:Conservative Versus Aggressive Discectomy
Brief Title: Conservative Versus Aggressive Discectomy for Primary Disc Herniation With Radiculopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Dongsheng Huang, MD., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zseyhds2
Record Dates: First submitted 2010-09-13; First posted 2010-09-17 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2007-08

CONDITIONS: Herniated Disc
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CS (Experimental): conservative discectomy
  Interventions: Procedure: conservative discectomy
- AS (Active Comparator)
  Interventions: Procedure: aggressive discectomy

INTERVENTIONS:
Procedure: conservative discectomy — a smaller incision with removal of the disc fragment with little invasion of the disc
  Arms: CS
Procedure: aggressive discectomy — a large open incision with aggressive removal of the disc fragments and curettage of the disc space
  Arms: AS

SUMMARY:
Summary: This is a prospective randomize study to compare conservative and aggressive discectomy for treatment of disc herniation with radiculopathy.

Study hypothesis: The investigators believe that conservative discectomy could preserve a higher disc space and has a better long-term outcomes.

DETAILED DESCRIPTION:
objectives:to compare the effect of two type surgery(conservative discectomy and aggressive discectomy)on disc herniation with radiculopathy after long-term follow-up.

methods:the patients who were confirmed suffer from disc herniation with radiculopathy and failed to nonsurgical treatment will be divided into two groups, and will be follow up 3~6 years for seeking the effect on disc space preservation and recurrent.

outcome measures:the rate of pain release and patients satisfaction were measured by SF-36,ODI,VAS,score post-OP. the height of disc was measured on X-ray film by the end point.

ELIGIBILITY:
Inclusion Criteria:

* Duration of symptoms: 6 or more weeks.
* Treatments tried: Non-steroidal anti-inflammatory medical therapy and physical therapy.
* Surgical screening: Persistent radicular pain provoked by moderate exercise, sitting, increased abdominal pressure, decreased mobility, list (scoliosis), straight leg raising.
* Tests: MRI to confirm diagnosis and level(s).

Exclusion Criteria:

* Previous lumbar spine surgery.
* Not a surgical candidate for any of these reasons: Overall health which makes spinal surgery too life-threatening to be an appropriate alternative, dramatic improvement with conservative care, or inability (for any reason) to undergo surgery within 6 months.
* Possible pregnancy.
* Active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer) is ineligible unless he or she has been treated with a curative intent AND there has been no clinical signs or symptoms of the malignancy for at least 5 years.
* Current fracture, infection, and/or deformity (greater than 15 degrees of lumbar scoliosis, using Cobb measure technique) of the spine.
* Age less than 18 years.
* Cauda Equina syndrome or progressive neurological deficit (usually requiring urgent surgery).
* Unavailability for follow-up (planning to move, no telephone, etc.) or inability to complete data surveys.
* Symptoms less than 6 weeks.
* Patient currently enrolled in any experimental "spine related" study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
patients satisfaction | 6 weeks after intervention
patients satisfaction | 3 months after intervention
patients satisfaction | 6 months after intervention
patients satisfaction | 1st year after intervention
patients satisfaction | 3rd year after intervention
patients satisfaction | 5th year after intervention

SECONDARY OUTCOMES:
recurrence rate of disc herniation | 6 weeks after operation
recurrence rate of disc herniation | 3 months after operation
recurrence rate of disc herniation | 6 months after operation
recurrence rate of disc herniation | 1st year after operation
recurrence rate of disc herniation | 3rd year after operation
recurrence rate of disc herniation | 5th year after operation
height of disc space | 6 weeks after operation
height of disc space | 3 months after operation
height of disc space | 6 months after operation
height of disc operation | 1st year after operation
height of disc space | 3rd year after operation
height of disc space | 5th year after operation

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Huang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen memorial hospital, Guangzhou, Guangdong, China